CLINICAL TRIAL: NCT01496651
Title: Nordic-Baltic-British Left Main Revascularization Study (NOBLE)
Brief Title: PCI vs. CABG in the Treatment of Unprotected Left Main Stenosis
Acronym: LeftMain/NOBLE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Evald Hoej Christiansen (Other)
Responsible Party: Sponsor-Investigator, Evald Hoej Christiansen, MD, DMSc, Aarhus University Hospital Skejby
Organization: Aarhus University Hospital Skejby (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LeftMain/NOBLE
Record Dates: First submitted 2011-12-19; First posted 2011-12-21 (Estimated); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Coronary Artery Disease
Keywords: Percutaneous coronary intervention; Coronary artery bypass graft operation; Left Main
MeSH Terms: conditions — Coronary Artery Disease | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Percutaneous coronary intervention (Active Comparator): Coronary Artery Bypass Grafting Versus Drug Eluting Stent Percutaneous Coronary Angioplasty in the Treatment of Unprotected Left Main Stenosis
  Interventions: Procedure: Percutaneous coronary intervention
- Coronary artery bypass graft operation (Active Comparator): Coronary Artery Bypass Grafting Versus Drug Eluting Stent Percutaneous Coronary Angioplasty in the Treatment of Unprotected Left Main Stenosis
  Interventions: Procedure: Coronary artery bypass graft operation

INTERVENTIONS:
Procedure: Percutaneous coronary intervention — PCI will be performed by the femoral or the transradial approach. In complex distal lesion anatomies, the use of 7-8F guiding catheters and the transfemoral approach may be recommended. Ostial and mid-shaft lesions will be treated with a single stent. For the treatment of distal bifurcation lesions crush, culotte, T-stenting, V-stenting or a single stent strategy may be used according the lesion morphology and the experience of the operator. However, based on the Nordic Bifurcation Studies the culotte technique seems to be associated with especially favorable angiographic and long-term clinical results in these large vessel size bifurcation lesions.
  There should be a low threshold for the use of high pressure post dilatation balloons. Generally, final kissing balloon dilatations are encouraged and mandatory when two-stent techniques are used. Intravascular ultrasound (IVUS) in mandatory pre and post stent placement.
  Other Names: PCI; PTCA
  Arms: Percutaneous coronary intervention
Procedure: Coronary artery bypass graft operation — Patients randomized to the CABG group for the treatment of LMCA stenosis are treated according to current clinical practice. Both off-pump and on-pump techniques can be used and the selection between the used methods is operator dependent. The left internal mammary artery will be used for the revascularization of the left anterior descending coronary artery, whenever feasible. For other lesion location, saphenous venous grafts, free arterial grafts or the right internal mammary artery may be used.
  Other Names: CABG
  Arms: Coronary artery bypass graft operation

SUMMARY:
Coronary Artery Bypass Grafting Versus Drug Eluting Stent Percutaneous Coronary Angioplasty in the Treatment of Unprotected Left Main Stenosis.

In a clinical, randomized, 5-year follow-up study to compare essential clinical outcome parameters in patients with unprotected left main (LMCA) disease, treated with coronary artery bypass grafting (CABG) versus percutaneous coronary intervention (PCI) using drug eluting stents (DES).

DES-PCI of unprotected LMCA disease is non-inferior to CABG concerning the 2-year rate of death, myocardial infarction, stroke or new revascularization and concerning the 5-year rate of death.

DETAILED DESCRIPTION:
Design:

Randomised open multicentre trial.

Patients:

Number 1,200

Randomisation:

PCI with DES vs CABG

Individuals for inclusion will be recruited among the patients referred to the participating centers for LMCA treatment. The patients will not be recruited by advertising and will receive no honorarium for participation.

Primary and secondary endpoints will be assessed by an independent endpoint committee (IEC). The endpoint committee will consist of experienced cardiac surgeons and cardiologists.

Follow-up All patients will be seen at the outpatient clinic of the participating centers after one month and after 1, 2 ,3 ,4 and 5 years. The outpatient visit may be substituted with a telephone contact and subsequent investigation and documentation of possible study events (MACCE). Finally, there will be a 10-year registry assessment of total mortality.

The index angiograms will be assessed by the QCA-laboratories at the Department of Cardiology, Aarhus University Hospital, Skejby, Denmark. The left main lesion and the non-left main lesions will be described and classified and a SYNTAX SCORE calculated.

The angiography obtained during the PCI-procedure will be used as index angiography. There should be at least two cine-runs before the procedure and after the procedure with the same angulations and proceeded by 0.1 mg intracoronary nitroglycerine (documented on the angiogram). The diagnostic/guiding catheter should be well visible, near the center of the angiogram and filled with dye. The index lesion should be well visible, near the centre of the angiogram and shown without foreshortening. There should be an angulation difference between the two baseline angiograms of at least 30 degrees. Between the pre and post angiograms all balloon inflations and stent implantations should be documented by short cine-runs.

Statistics and data management:

The statistical analyses will be performed at the Department of Clinical Epidemiology, Aarhus University Hospital.

Analysis population:

The results will be analyzed according to the intention-to-treat principle, i.e. patients randomized to a certain group will be followed and assessed irrespectively of the actual treatment. Protocol violations will be noted and the responsible centers notified.

Sample size calculations:

Primary endpoint of 2-year MACCE Sample size calculation is based on the combined primary endpoint of death, stroke, non-index treatment related MI and new revascularization (PCI or CABG) after 2 years.

The study is planned as a non-inferiority study, where an experimental treatment of a disease (E, here PCI) is compared to a standard treatment (S, here CABG). E is not allowed to be more than clinically insignificantly inferior to S to be declared non-inferior. Calculations are based on the following:

* mean follow-up time 24 months
* all event curves are exponential
* zero dropout
* randomization into 2 equally sized groups
* α = 0.05 (one-sided)
* 1- β (power) = 80% The non-inferiority limit is based on a 12 months MACCE rate of 12% in the CABG and 16% in the PCI group (the SYNTAX study). With exponential event curves (S(t)=exp(-λ*t)) this corresponds to a hazard ratio of 1.36, PCI versus CABG, and, with t in months, λ=0.0107 in the CABG group. In continuation if this, the present study uses hazard ratio 1.35, E versus S, as limit for non-inferiority, and λ=0.011 to describe MACCE in the CABG group. These figures correspond to a 24-month MACCE rate of 30% and 23% in the PCI and CABG group, respectively.

The above preconditions and assumptions result in a necessary number of patients in each randomization group of 593 (and a total number of events - in both groups - of 275). Consequently, 1,186 patients should be randomized.

By including 600 patients in each group, possible dropouts before follow-up and treatment estimation errors are accounted for.

Data management The study is reported to Danish Data Protection Agency, and the agency's guidelines for data management will be followed. Dedicated case record forms will be used and faxed to PCI research, Cardiac Cath. Lab., Aarhus University Hospital, Skejby, 8200 Aarhus N, Denmark. Data will be stored in an Access database and double data entry will be used as quality control. There will be a log of accesses and attempt of accesses. Back-up data and original data will be encrypted.

Monitoring of the study:

The study will be monitored according to the GCP rules by independent professionals. During the study period, monitors will have regular contact to the participating departments to ensure that the trial is conducted in compliance with the protocol, GCP and applicable regulatory requirements.

The monitors will ensure that the used products are all right and will review source documents for verification of consistency with the data recorded in the CRFs. The monitors will also provide information and support to the investigator(s).

Investigators and other responsible personnel must be available during the monitoring visits, audits and inspections and should devote sufficient time to these processes.

The investigator should provide a CV or equivalent documentation of suitability to be responsible for the trial. All investigators and other responsible personnel should be listed together with their function in the trial on the signature list.

Publication:

Results, positive as well as negative, will be published in an international cardiovascular journal. Publication and author issues will be decided by the steering committee on basis of general involvement in the study (drafting of protocol, core lab. function, endpoint committee membership, etc.) and on number of included patients. Thus, the sequence of authors will be determined by the inclusions rates of the participating centres and the most including centre will be offered the position as first author.

ELIGIBILITY:
Inclusion Criteria:

* Stable, unstable angina pectoris or ACS.
* Significant lesion* of LMCA ostium, mid-shaft and/or bifurcation and with no more than three additional non-complex** PCI lesions.
* Patient eligible to be treated by CABG and by PCI
* Signed informed consent. *Visually assessed diameter stenosis >50% or fractional flow reserve <0.80. **Length <25 mm, non-CTO, non-2-stent bifurcation, non-calcified and non-tortuous vessel morphology coronary lesion.

Exclusion Criteria:

* ST-elevation infarction within 24 hours.
* CABG clearly better treatment option (LMCA stenosis and >3, or complex** additional coronary lesions)
* Patient is in too high risk for CABG.
* Expected survival <1 year.
* Allergy to aspirin, clopidogrel or ticlopidine.
* Allergy to Biolimus. **Length >25 mm, CTO, 2-stent bifurcation, calcified or tortuous vessel morphology coronary lesion.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1201 (Actual)
Dates: Start 2008-11-06 (Actual); Primary Completion 2015-01-22 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Combined endpoint of death, stroke, non-index treatment related MI and new revascularization (PCI or CABG) | From date of first randomisation until a total number of 275 events is reached (or max 5 years).

SECONDARY OUTCOMES:
Combined endpoint of death, stroke and non-index treatment related MI | 30 days, yearly through 5 years and when a total number of 275 events is reached.
Individual endpoints of death, stroke and non-index treatment related MI | 30 days, yearly through 5 years and when a total number of 275 events is reached.
All cause mortality | 10 years
New revascularization by CABG or PCI | 30 days, yearly through 5 years and when a total number of 275 events is reached.
Death | 30 days, yearly through 5 years and when a total number of 275 events is reached.
Definite stent thrombosis/symptomatic graft occlusion | 30 days, yearly through 5 years and when a total number of 275 events is reached.
CCS angina score | 30 days, yearly through 5 years and when a total number of 275 events is reached.
NYHA functional class | 30 days, yearly through 5 years and when a total number of 275 events is reached.
Duration of admission for index treatment | Baseline
Syntax score | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Evald H Christiansen, MD, Principal Investigator — Aarhus University Hospital Skejby
Locations (1):
- Aarhus University Hospital, Skejby, Aarhus N, Denmark

REFERENCES:
- [Derived] Gaba P, Christiansen EH, Nielsen PH, Murphy SA, O'Gara PT, Smith PK, Serruys PW, Kappetein AP, Park SJ, Park DW, Stone GW, Sabik JF, Sabatine MS, Holm NR, Bergmark BA. Percutaneous Coronary Intervention vs Coronary Artery Bypass Graft Surgery for Left Main Disease in Patients With and Without Acute Coronary Syndromes: A Pooled Analysis of 4 Randomized Clinical Trials. JAMA Cardiol. 2023 Jul 1;8(7):631-639. doi: 10.1001/jamacardio.2023.1177. PMID 37256598
- [Derived] Steigen T, Holm NR, Myrmel T, Endresen PC, Trovik T, Makikallio T, Lindsay M, Spence MS, Erglis A, Menown IBA, Kumsars I, Kellerth T, Davidavicius G, Linder R, Anttila V, Juul Hune Mogensen L, Hostrup Nielsen P, Graham ANJ, Hildick-Smith D, Thuesen L, Christiansen EH; NOBLE Study Investigators. Age-Stratified Outcome in Treatment of Left Main Coronary Artery Stenosis: A NOBLE Trial Substudy. Cardiology. 2021;146(4):409-418. doi: 10.1159/000515376. Epub 2021 Apr 13. PMID 33849035
- [Derived] Holm NR, Makikallio T, Lindsay MM, Spence MS, Erglis A, Menown IBA, Trovik T, Kellerth T, Kalinauskas G, Mogensen LJH, Nielsen PH, Niemela M, Lassen JF, Oldroyd K, Berg G, Stradins P, Walsh SJ, Graham ANJ, Endresen PC, Frobert O, Trivedi U, Anttila V, Hildick-Smith D, Thuesen L, Christiansen EH; NOBLE investigators. Percutaneous coronary angioplasty versus coronary artery bypass grafting in the treatment of unprotected left main stenosis: updated 5-year outcomes from the randomised, non-inferiority NOBLE trial. Lancet. 2020 Jan 18;395(10219):191-199. doi: 10.1016/S0140-6736(19)32972-1. Epub 2019 Dec 23. PMID 31879028
- [Derived] Makikallio T, Holm NR, Lindsay M, Spence MS, Erglis A, Menown IB, Trovik T, Eskola M, Romppanen H, Kellerth T, Ravkilde J, Jensen LO, Kalinauskas G, Linder RB, Pentikainen M, Hervold A, Banning A, Zaman A, Cotton J, Eriksen E, Margus S, Sorensen HT, Nielsen PH, Niemela M, Kervinen K, Lassen JF, Maeng M, Oldroyd K, Berg G, Walsh SJ, Hanratty CG, Kumsars I, Stradins P, Steigen TK, Frobert O, Graham AN, Endresen PC, Corbascio M, Kajander O, Trivedi U, Hartikainen J, Anttila V, Hildick-Smith D, Thuesen L, Christiansen EH; NOBLE study investigators. Percutaneous coronary angioplasty versus coronary artery bypass grafting in treatment of unprotected left main stenosis (NOBLE): a prospective, randomised, open-label, non-inferiority trial. Lancet. 2016 Dec 3;388(10061):2743-2752. doi: 10.1016/S0140-6736(16)32052-9. Epub 2016 Oct 31. PMID 27810312